CLINICAL TRIAL: NCT04536324
Title: The Absorption Rate of Subcutaneous Infused Fluid in Both Acutely Ill and Healthy Older Adults
Brief Title: The Absorption Rate of Subcutaneous Infused Fluid
Acronym: ABSU
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Mathias Aalkjær Brix Danielsen, MD, Aalborg University Hospital
Other Study IDs: N-20200010
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Aged, 75 and Over; Aged; Hypodermoclysis; Fluid Therapy; Dehydration
Keywords: Dehydration; Fluid therapy; Hypodermoclysis; Geriatric; Sodium Pertechnetate Tc 99m
MeSH Terms: conditions — Dehydration | interventions — Hypodermoclysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Subcutaneous parenteral hydration — Patients will twice receive a subcutaneous infusion of 250 ml isotonic sodium chloride (NaCl) with 30 MBq Tc-99m pertechnetate mixed in. The patients will receive the first infusion during admission to our geriatric ward (when they are acutely ill) and the second infusion approximately 8 weeks after discharge when they are no longer acutely ill. The subcutaneous access will be placed on the abdomen in the lower left or right quadrant.
  Other Names: Hypodermoclysis

SUMMARY:
The purpose of the study is to examine the rate of absorption of subcutaneous infused fluid in older adults when acutely ill compared to when they are not acutely ill.

DETAILED DESCRIPTION:
Dehydration is a common condition in older adults. When oral hydration is insufficient there is a need for parenteral hydration. Subcutaneous infused fluid or hypodermoclysis is a method for parenteral hydration. This method is used to treat older adults with mild to moderate dehydration or at risk of dehydration. Despite that, this method is used in older adults who are acutely ill we have a very limited understanding of the absorption time and thereby when the infused fluid is available in the circulatory system. This study aims to compare the absorption time in older adults who are acutely ill with when they are not acutely ill. Furthermore, this study aims to describe how fast the subcutaneous infused fluid is absorbed from the subcutaneous space and subsequently when it is available in the circulatory system where it has its effect.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Hospitalized for an acute illness

Exclusion Criteria:

* Severe limitation on fluids
* Risk of acute deterioration of illness
* Requiring constant care
* Short life expectancy

Ages: 75 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to the local geriatric ward will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
The difference in the absorption rate between acutely ill and not acutely ill. | 8 weeks after discharge
  We will compare the absorptions rate of subcutaneous infused fluid when the patients are acutely ill (during admission) and when they are not acutely ill (8 weeks after discharge).

SECONDARY OUTCOMES:
The absorption rate of subcutaneous infused fluid by count over the infusion site | We will count the activity from the start of infusions until 2 hours after all of the 250 ml have been infused.
  From the start of the infusion, we will count the activity with a gamma detector (CAPTUS® 3000, Capintec Inc. Pittsburgh). From this data, we will estimate the absorption rate of the subcutaneous infused fluid.
The absorption rate of subcutaneous infused fluid by count in the thyroid or by count in blood samples. | We will count the activity from the start of infusions until 2 hours after all of the 250 ml have been infused.
  We will also assess the absorption of the subcutaneously infused fluid by registering the activity in the patients' thyroid gland. If the activity in the thyroid is to low to properly register we will measure the activity in the patients' blood samples.
  We will use a gamma detector (CAPTUS® 3000, Capintec Inc. Pittsburgh) to count the activity in both the thyroid and blood samples.
The correlation between s-albumin and absorption time. | We will count the activity from the start of infusions until 2 hours after all of the 250 ml have been infused.
  As albumin is an important contributor of the osmotic pressure of serum we will in investigate if there is a correlation between the level of s-albumin and absorption rate.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias B Danielsen, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification. Data sets will only be shared when the anonymity of included participants can be insured.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Beginning 6 months and ending 5 years following article publication.
Access Criteria: The dataset will be shared upon reasonable request.

REFERENCES:
- [Derived] Danielsen MB, Jodal L, Riis J, Karmisholt JS, Valdorsson O, Jorgensen MG, Andersen S. Absorption rate of subcutaneously infused fluid in ill multimorbid older patients. PLoS One. 2022 Oct 10;17(10):e0275783. doi: 10.1371/journal.pone.0275783. eCollection 2022. PMID 36215232